CLINICAL TRIAL: NCT02092597
Title: Safety Evaluation of Adverse Reactions in Diabetes
Acronym: SAFEGUARD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Martin Haluzik, Professor, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEALTH-282521-CUNI
Record Dates: First submitted 2014-03-18; First posted 2014-03-20 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide; Linagliptin; Gliclazide

ARMS (3):
- GLP-1 agonist (Active Comparator): Exenatide 5 ug s.c. bid for the 1st month, 10 ug s.c. bid for the next 2 months
  Interventions: Drug: Exenatide
- DPP-4 inhibitor (Active Comparator): Linagliptin 5 mg tbl qd for 3 months
  Interventions: Drug: Linagliptin
- Sulfonylurea derivate (Active Comparator): Gliclazid 30 mg tbl qd for 3 months
  Interventions: Drug: Gliclazide

INTERVENTIONS:
Drug: Exenatide
  Arms: GLP-1 agonist
Drug: Linagliptin
  Arms: DPP-4 inhibitor
Drug: Gliclazide
  Arms: Sulfonylurea derivate

SUMMARY:
The purpose of this study is to assess the effects of incretin-based antidiabetic therapies (DPP-4 inhibitors and GLP-1 agonists) on cardiovascular, gastrointestinal and renal system and to detail the mechanisms underlying their action in these systems.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Metformin monotherapy - stable dose during last 3 months
* HbA1C 48-75 mmol/mol (IFCC)
* BMI 25-40 kg/m2
* Age 35-70 years (women postmenopausal)
* Use of ACE inhibitors or ATII receptor blockers for at least 3 months before enrollment

Exclusion Criteria:

* eGFR<30 ml/min/1.73m2 (MDRD)
* Treatment with incretin mimetics during 3 months before enrollment
* Chronic insulin therapy
* Chronic use of loop diuretics, glucocorticoids, NSAID, immune suppressants, antimicrobial agents, chemotherapeutics, bile acid sequestrants (colestyramin, colesevelam)
* History of pancreatic disease or impaired pancreatic function (defined as the need to use pancreatic enzymes)
* Active liver disease or a 3-fold elevation of liver transaminases (ALT, AST)
* Active malignancy
* History of severe cardiovascular disease including acute coronary syndrome, stroke or transient ischemic neurologic disorder during previous 6 months, atrial fibrillation or other arrhythmia requiring chronic antiarrhythmic medication, chronic heart failure (New York Heart Association grade III/IV)
* History of alcohol abuse, defined as >4 units of alcohol/day (32 g or 40 ml of 100% alcohol)
* History of allergy for GLP-1 receptor agonists or DPP-4 inhibitors
* Any disease that could interfere with study procedures (e.g. decreased mobility, mental incapacity)
* Inability to give informed consent

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Heart rate | 90 days after treatment initiation
Gastric evacuation velocity | 90 days after treatment initiation
Blood pressure | 90 days after treatment initiation
Left ventricular ejection fraction | 90 days after treatment initiation
Intimomedial thickness | 90 days after treatment initiation
Pulse wave velocity | 90 days after treatment initiation
Glomerular filtration rate | 90 days after treatment initiation
Tubular function | 90 days after treatment initiation
KIM-1 | 90 days after treatment initiation
  Marker of renal damage
Exocrine pancreas function | 90 days after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Martin Haluzik, MD DSc, Principal Investigator — 3rd Department of Medicine, General University Hospital and Charles University 1st Faculty of Medicine
Locations (1):
- General University Hospital, Prague, Czechia